CLINICAL TRIAL: NCT03941249
Title: Blood Biomarkers of Metabolic Processes (Metabolomics) and Brain Derived Proteins in Stroke Patients.
Brief Title: Blod Biomarkers for Stroke
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Helle Klingenberg Iversen, MD, DmSc (Other)
Responsible Party: Sponsor-Investigator, Helle Klingenberg Iversen, MD, DmSc, MD, DmSc, head of the stroke unit, Glostrup University Hospital, Copenhagen
Organization: Glostrup University Hospital, Copenhagen (Other)
Other Study IDs: H-15021321
Record Dates: First submitted 2017-12-04; First posted 2019-05-07 (Actual); Last update posted 2022-03-29 (Actual); Status verified 2022-03

CONDITIONS: Stroke
Keywords: Metabolomics; Tau; Ischemic stroke; Hemorrhagic stroke
MeSH Terms: conditions — Stroke; Pick Disease of the Brain; Ischemic Stroke; Hemorrhagic Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Biospecimen Retention: Samples With DNA — Blodsampels
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of the project is to investigate specific markers in blood samples from patients with stroke (ischemic or hemorrhagic). This could hopefully help in the early diagnostic to separate patients with ischemic stroke from those with hemorrhagic stroke as treatment are different and patients need to come quickly to the correct treatment site.

DETAILED DESCRIPTION:
Approximately 12,000 Danes suffer a stroke each year with major consequences for those affected, their relatives and society in general. Rapid diagnosis and treatment mean less brain damage and thus less risk of late sequelae. A marker in the blood that is specific for stroke could result in faster diagnose and thereby treatment. Until now, no such marker has been found, but measurement of the so-called metabolomics and different fragments of brain proteins like Tau has shown promising results. Currently, metabolomics has only been studied in two other projects in stroke patients, and the results were not complete and a subtype of Tau (Tau-C) has been shown to be related to brain damage after ice hockey, but this is not studied in stroke patients, so there is a need for more studies.

In this project different fragments of brain proteins and the so-called metabolomics in the blood, which are small residues from the biological processes that take place in the body, such as fat and sugar incineration, will be studied.

The project is based on blood samples from a biobank that has been established in connection with previous projects in the Stroke Unit, Neurological Clinic, Rigshospitalet, Glostrup. All subjects have given written consent to give blood for future research.

Fifty microliters of blood from each participant will be analyzed by so-called mass spectroscopy, a well-researched method and performed in a recognized laboratory using known libraries and databases of metabolites for the determination and ongoing quality control. In addition, 250 microliters of serum will be analyzed by Elisa to detect brain proteins like Tau and Brevican.

The metabolomic profile and the brain proteins is compared to the information we have about the participants, namely:

* If they had ischemic or hemorrhagic stroke or if it is a healthy control person
* The extent of brain damage; partly measured by the brain scan and partly from the patient's symptoms
* The cause of the stroke

ELIGIBILITY:
Inclusion Criteria:

* Clinical stroke

Exclusion Criteria:

* Glasgow Coma Scale (GCS) < 15
* Non communicating patients e.g. aphasia (incompetent patients)
* Unable to cooperate to the physical examinations
* Pregnancy or nursing mothers
* If the investigators find the study participant unfit to conduct the investigations

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Stroke patients admitted to the acute stroke unit at Rigshospitalet, Glostrup. Healthy volunteers.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2017-11-01 (Actual); Primary Completion 2023-04-30 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Ischemic or hemorrhagic stroke | Within 7 days
  We hope to find a method to differentiate between ischemic and hemorrhagic stroke.

SECONDARY OUTCOMES:
The extend of the brain damage | Within 7 days
  The relation between the biomarkers and brain damage measured by MRI.
The extend of the physical damage | Within 7 days
  The relation between the biomarkers and brain damage measured by NIHSS.
Etiology of stroke | Within 7 days
  The relation between the biomarkers and stroke etiology measured by the TOAST criteria.
Stroke patient or healthy subject | Within 7 days
  The relation between the biomarkers and healthy subjects.

CONTACTS AND LOCATIONS:
Overall Officials: Helle K Iversen, MD, DMSc, Principal Investigator — Department of clinical stroke research, Neurological department, Rigshospitalet, Glostrup
Locations (1):
- Department of clinical stroke research, department of neurology, Glostrup Hospital, Glostrup Municipality, Denmark